CLINICAL TRIAL: NCT00868790
Title: A Phase IIa, Multicenter, Randomized, Placebo- and Active-Comparator Controlled, Cross-Over Clinical Trial to Study the Safety and Efficacy of MK-3577 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: A Study of the Safety and Efficacy of MK-3577 in Participants With Type 2 Diabetes Mellitus (MK-3577-009)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Upon interim analysis, sufficient data was accrued to assess study hypotheses.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3577-009; 2009_564 (Other: Merck Registration Number); CTRI/2009/091/000614 (Registry Identifier: CTRI)
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) (Experimental): Participants were to receive oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4. Domiciled participants were also to receive placebo to metformin during Period 1 and Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Placebo to Metformin
- MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) (Experimental): Participants were to receive oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4. Domiciled participants were also to receive placebo to metformin during Period 1 and Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Placebo to Metformin
- MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) (Experimental): Participants were to receive oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed MK- 3577 25 mg BID for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) (Experimental): Participants were to receive oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) (Experimental): Participants were to receive oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 25 mg BID for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) (Experimental): Participants were to receive oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) (Experimental): Participants were to receive oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) (Experimental): Participants were to receive oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) (Experimental): Participants were to receive oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during period 4. Domiciled participants were also to receive placebo to metformin during Period 1 and Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Placebo to Metformin
- MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) (Experimental): Participants were to receive oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by MK-3577 25 mg BID for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) (Experimental): Participants were to receive oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4. Domiciled participants were also to receive placebo to metformin during Period 1 and Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Placebo to Metformin
- MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) (Experimental): Participants were to receive oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577
- PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) (Experimental): Domiciled participants were to receive oral treatment with dose-matched placebo to metformin (METF) for 4 weeks during Period 1, followed by metformin 1000 mg BID for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4. Participants in this arm were administered metformin placebo during Period 1 and active metformin during Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Metformin; Drug: Placebo to Metformin
- METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14) (Experimental): Domiciled participants were to receive oral treatment with metformin 1000 mg BID for 4 weeks during Period 1, followed by dose-matched placebo to metformin for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4. Participants in this arm were administered active metformin during Period 1 and metformin placebo during Period 2.
  Interventions: Drug: MK-3577; Drug: Placebo to MK-3577; Drug: Metformin; Drug: Placebo to Metformin

INTERVENTIONS:
Drug: MK-3577 — MK-3577 oral tablets totaling 6 mg in the evening (PM), 10 mg in the morning (AM), or 25 mg twice daily (BID) depending upon randomization, administered during a 4 week treatment period.
Drug: Placebo to MK-3577 — Dose-matched placebo tablets to MK-3577 administered during a 4 week treatment period
Drug: Metformin — Two 500 mg tablets of metformin were administered twice daily (2000 mg total daily dose) to domiciled participants during a 4 week treatment period.
  Arms: METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14); PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13)
Drug: Placebo to Metformin — Two placebo tablets to metformin were administered twice daily (2000 mg total daily dose) to domiciled participants during a 4 week treatment period.
  Arms: METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14); MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2); MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11); PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13); PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1); PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9)

SUMMARY:
This study assessed the safety and efficacy of MK-3577. The primary efficacy hypothesis was that, after 4 weeks of treatment, either the morning (AM) administration or the evening (PM) administration of MK-3577 provides superior reduction of 24-hour weighted mean glucose (WMG) levels compared to placebo (PLA). The primary safety hypothesis was that MK-3577 is well tolerated compared to placebo.

DETAILED DESCRIPTION:
This was a 4-period/5-treatment crossover study. Each period was 4 weeks. The 5 treatments consisted of MK-3577 10 mg once daily (QD) in the AM, MK-3577 6 mg QD in the evening (PM), MK-3577 25 mg twice daily (BID), metformin 1000 mg BID, and placebo to MK-3577/placebo to metformin. Participants were to be randomized to one of 14 treatment sequence arms. A subset of participants in each group was to domicile (stay overnight) at selected clinical sites at Baseline, Week 4 (end of Period 1), and Week 8 (end of Period 2) to undergo 24-hr blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Participant has type 2 diabetes
* Participant is either not taking antihyperglycemic medications for the last 10 weeks OR is taking a single oral antihyperglycemic medication (but not a Peroxisome Proliferator-Activated Receptor gamma [PPARg] agonist) OR is taking a low-dose combination oral antihyperglycemic medication (not a PPARg agonist) at dose less than or equal to 50% of the maximum dose
* Female participant is unable to have children

Exclusion Criteria:

* Participant has a history of type 1 diabetes or ketoacidosis
* Participant has been treated with a PPARg agonist in the last 12 weeks
* Participant has been treated with insulin in the last 12 weeks
* Participant has had prescription lipid-modifying drug therapy in the last 12 weeks
* Participant has a history of coronary artery disease
* Participant has had a stroke or transient ischemic attack
* Participant has congestive heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2010-07-12 (Actual); Study Completion 2010-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=3577-009&kw=3577-009&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 118 participants were randomized to one of 14 treatment sequence arms on this cross-over study. Each participant received 4 out of 5 treatments over 4 treatment periods. Before randomization, participants who had prior antihyperglycemic agent (AHA) treatment had a 4-week AHA wash-off, and all participants had a 2-week placebo run-in.
Groups:
- PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1): Participants received oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4. Domiciled participants also received placebo to metformin during Period 1 and Period 2.
- MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2): Participants received oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4. Domiciled participants also received placebo to metformin during Period 1 and Period 2.
- MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3): Participants received oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed MK- 3577 25 mg BID for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4.
- MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4): Participants received oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
- PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5): Participants received oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 25 mg BID for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4.
- MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6): Participants received oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4.
- MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7): Participants received oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
- MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8): Participants received oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4.
- PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9): Participants received oral treatment with dose-matched placebo to MK-3577 for 4 weeks during Period 1, followed by MK-3577 6 mg QD PM for 4 weeks during Period 2, followed by MK-3577 25 mg BID for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during period 4. Domiciled participants also received placebo to metformin during Period 1 and Period 2.
- MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10): Participants received oral treatment with MK-3577 10 mg QD AM for 4 weeks during Period 1, followed by MK-3577 25 mg BID for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 4.
- MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11): Participants received oral treatment with MK-3577 6 mg QD PM for 4 weeks during Period 1, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 25 mg BID for 4 weeks during Period 4. Domiciled participants also received placebo to metformin during Period 1 and Period 2.
- MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12): Participants received oral treatment with MK-3577 25 mg BID for 4 weeks during Period 1, followed by MK-3577 10 mg QD AM for 4 weeks during Period 2, followed by dose-matched placebo to MK-3577 for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4.
- PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13): Domiciled participants received oral treatment with dose-matched placebo to metformin (METF) for 4 weeks during Period 1, followed by metformin 1000 mg BID for 4 weeks during Period 2, followed by MK-3577 10 mg QD AM for 4 weeks during Period 3, followed by MK-3577 6 mg QD PM for 4 weeks during Period 4. Participants in this arm were administered metformin placebo during Period 1 and active metformin during Period 2.
- METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14): Domiciled participants received oral treatment with metformin 1000 mg BID for 4 weeks during Period 1, followed by dose-matched placebo to metformin for 4 weeks during Period 2, followed by MK-3577 6 mg QD PM for 4 weeks during Period 3, followed by MK-3577 10 mg QD AM for 4 weeks during Period 4. Participants in this arm were administered active metformin during Period 1 and metformin placebo during Period 2.
Period: Period 1
Arm/Group | PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) | MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) | MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) | MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) | PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) | MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) | MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) | MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) | PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) | MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) | MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) | MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) | PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) | METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14)
Started | 11 | 8 | 4 | 4 | 19 | 3 | 4 | 20 | 11 | 3 | 9 | 4 | 7 | 11
Completed | 9 | 7 | 4 | 4 | 18 | 2 | 4 | 17 | 10 | 3 | 9 | 4 | 7 | 9
Not Completed | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Abnormal Triglycerides | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) | MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) | MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) | MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) | PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) | MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) | MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) | MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) | PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) | MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) | MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) | MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) | PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) | METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14)
Started | 9 | 7 | 4 | 4 | 18 | 2 | 4 | 17 | 10 | 3 | 9 | 4 | 7 | 9
Completed | 9 | 6 | 4 | 4 | 18 | 1 | 4 | 17 | 8 | 3 | 9 | 4 | 7 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) | MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) | MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) | MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) | PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) | MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) | MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) | MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) | PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) | MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) | MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) | MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) | PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) | METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14)
Started | 9 | 6 | 4 | 4 | 18 | 1 | 4 | 17 | 8 | 3 | 9 | 4 | 7 | 8
Completed | 9 | 6 | 4 | 3 | 18 | 1 | 4 | 17 | 8 | 2 | 8 | 4 | 7 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) | MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) | MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) | MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) | PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) | MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) | MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) | MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) | PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) | MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) | MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) | MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) | PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) | METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14)
Started | 9 | 6 | 4 | 3 | 18 | 1 | 4 | 17 | 8 | 2 | 8 | 4 | 7 | 8
Completed | 7 | 6 | 3 (One non-completion due to abnormal alanine aminotransferase/aspartate aminotransferase (ALT/AST)) | 3 | 18 | 1 | 4 | 14 | 6 | 2 | 5 | 3 | 6 | 7
Not Completed | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 1
Not completed — Abnormal ALT/AST | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post-study
Arm/Group | PLA→MK-3577 QD AM→MK-3577 QD PM→MK-3577 BID (Arm 1) | MK-3577 QD AM→PLA→MK-3577 BID→MK-3577 QD PM (Arm 2) | MK-3577 QD PM→MK-3577 BID→PLA→MK-3577 QD AM (Arm 3) | MK-3577 BID→MK-3577 QD PM→MK-3577 QD AM→PLA (Arm 4) | PLA→MK-3577 BID→MK-3577 QD AM→MK-3577 QD PM (Arm 5) | MK-3577 QD AM→MK-3577 QD PM→PLA→MK-3577 BID (Arm 6) | MK-3577 QD PM→MK-3577 QD AM→MK-3577 BID→PLA (Arm 7) | MK-3577 BID→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 8) | PLA→MK-3577 QD PM→MK-3577 BID→MK-3577 QD AM (Arm 9) | MK-3577 QD AM→MK-3577 BID→MK-3577 QD PM→PLA (Arm 10) | MK-3577 QD PM→PLA→MK-3577 QD AM→MK-3577 BID (Arm 11) | MK-3577 BID→MK-3577 QD AM→PLA→MK-3577 QD PM (Arm 12) | PLA→METF→MK-3577 QD AM→MK-3577 QD PM (Arm 13) | METF→PLA→MK-3577 QD PM→MK-3577 QD AM (Arm 14)
Started | 7 | 6 | 3 | 3 | 18 | 1 | 4 | 14 | 6 | 2 | 5 | 3 | 6 | 7
Completed | 7 | 6 | 3 | 3 | 17 | 1 | 4 | 12 | 6 | 1 | 5 | 3 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Excluded Medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who took at least one dose of study treatment
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) After 4-Week Treatment in Weighted Mean Glucose (WMG)
Description: The primary efficacy outcome in this study was the assessment of 24-hour weighted mean glucose (WMG) levels for domiciled participants after 4-week treatment (Periods 1 and 2 only). At selected study sites, a subset of participants domiciled (stayed) overnight and underwent 24-hour blood sampling at the Week 0 Visit (Baseline), Week 4 Visit (end of Period 1), and Week 8 Visit (end of Period 2). Domiciled participants were not expected to follow a weight-maintaining diet while receiving standard meals from a dietician or licensed healthcare professional. WMG was calculated as the weighted average value of the glucose from the 24-hour blood sample (for Baseline, Week 4, and Week 8) and analyzed using a Longitudinal Data Analysis (LDA) model. Results were expressed as the change from baseline after 4-week treatment in 24-hour WMG.
Time Frame: Week 0 Visit (Baseline), Week 4 Visit, Week 8 Visit
Population: All randomized domiciled participants receiving ≥1 dose of therapy and having 24-hour WMG measurement either at BL or end of Treatment Period 1 or 2. Number of Participants Analyzed=number of participants included in LDA model. Participants in MK-3577 25 mg BID group did not undergo 24-hour glucose sampling and were not analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo (PLA): Participants received dose-matched placebo tablets to MK-3577 (10 mg, 6 mg, 25 mg) and metformin, depending upon randomization, for 4 weeks.
- MK-3577 AM: Domiciled participants received MK-3577 10 mg orally every day (QD) in the morning (AM) for 4 weeks
- MK-3577 PM: Domiciled participants received MK-3577 6 mg orally QD in the evening (PM) for 4 weeks.
- MK-3577 BID: Domiciled participants received MK-3577 25 mg orally twice daily (BID) for 4 weeks.
- METF BID: Domiciled participants received metformin 1000 mg orally BID 4 weeks (received during Period 1 or 2 only).
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 38 | 10 | 11 | 0 | 15
mg/dL | -1.6 (4.1) | -18.8 (6.8) | -25.0 (6.7) |  | -36.5 (6.1)
Statistical Analysis 1: Comparison: Placebo (PLA) vs MK-3577 AM; Analysis based on an LDA model including terms for treatment, period, the interaction of treatment by period, prior antihyperglycemic therapy status (yes/no), and randomization stratum (participation in domiciled visits [yes/no]). The LDA-model test was conducted at alpha level=0.10 (two sided); Test type: Superiority or Other; p = 0.013, LDA Model; Between-group difference (MK-3577-placebo) of LSM changes from BL to a given time point and 90% confidence intervals were estimated from LDA model; Least Squares Mean (LSM) Difference = -17.2, 90% CI 2-sided [-28.3 to -6.1]
Statistical Analysis 2: Comparison: Placebo (PLA) vs MK-3577 PM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -23.4, 90% CI 2-sided [-34.5 to -12.4]
Statistical Analysis 3: Comparison: Placebo (PLA) vs METF BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; Between-group difference (metformin-placebo) of LSM changes from BL to a given time point and 90% confidence intervals were estimated from LDA model; LSM Difference = -34.9, 95% CI 2-sided [-44.8 to -25.0]

2. Secondary Outcome: Change From Baseline (BL) After 4-Week Treatment in Fasting Plasma Glucose (FPG)
Description: Fasting blood samples were obtained during study site visits at Baseline (Week 0 Visit) and Week 4 of each treatment period (Week 4 Visit, Week 8 Visit, Week 12 Visit, Week 16 Visit). Participants were counseled to fast (no food or drink except water and non-study medications, as directed) for at least 12 hours prior to all study visits. FPG was analyzed using an LDA model, and change from baseline (Week 0) after 4-week treatment in FPG was reported.
Time Frame: Week 0 Visit (Baseline), Week 4 Visit, Week 8 Visit, Week 12 Visit, Week 16 Visit
Population: All randomized participants receiving ≥1 dose of therapy and having FPG measurement either at BL or end of Treatment Period. Number of Participants Analyzed=number of participants included in the LDA model.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- MK-3577 AM: Participants received MK-3577 10 mg orally every day (QD) in the morning (AM) for 4 weeks.
- MK-3577 PM: Participants received MK-3577 6 mg orally QD in the evening (PM) for 4 weeks.
- MK-3577 BID: Participants received MK-3577 25 mg orally twice daily (BID) for 4 weeks.
- METF BID: Domiciled participants received metformin 1000 mg orally BID for 4 weeks (received during Period 1 or 2 only).
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 104 | 100 | 98 | 86 | 18
mg/dL | 4.3 (3.8) [-17.5 to -5.4] | -7.2 (3.5) [-27.8 to -15.8] | -17.5 (3.5) [-42.0 to -30.0] | -31.7 (3.5) [-30.0 to -10.1] | -14.4 (6.2)
Statistical Analysis 1: Comparison: Placebo (PLA) vs MK-3577 AM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -11.5, 90% CI 2-sided [-17.5 to -5.4]
Statistical Analysis 2: Comparison: Placebo (PLA) vs MK-3577 PM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -21.8, 90% CI 2-sided [-27.8 to -15.8]
Statistical Analysis 3: Comparison: Placebo (PLA) vs MK-3577 BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -36.0, 90% CI 2-sided [-42.0 to -30.0]
Statistical Analysis 4: Comparison: Placebo (PLA) vs METF BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, LDA Model; [statistical method as in outcome 1, analysis 3]; LSM Difference = -20.0, 90% CI 2-sided [-30.0 to -10.1]

3. Secondary Outcome: Change From BL After 4-Week Treatment in 2-hour Post-Meal Glucose (PMG) Levels
Description: Two-hour PMG was analyzed in both non-domiciled and domiciled participants. Non-domiciled participants completed a 3-point meal tolerance test (MTT) at Week 0 (Baseline) and Week 4 Visits of Treatment Period 1. Participants completed 12-hr fasting prior to the Week 0 (Baseline) and Week-4 clinic visits. Fasting blood samples were obtained at the beginning of these clinic visits, after which participants consumed a standardized meal (1 nutrition bar and 1 can of nutrition drink), and then completed the MTT, in which plasma glucose was measured at 30 min and 120 min (2 hr) post-meal. The 2-hr PMG data also include data from domiciled participants, based on 2-hr post-morning meal glucose levels in the 24-hr blood glucose sample at the Week 4 and Week 8 Visits. The 2-hour PMG was analyzed using an LDA model, and change from baseline (Week 0) after 4-week treatment in 2-hour PMG was reported.
Time Frame: Week 0 Visit (Baseline), Week 4 Visit, Week 8 visit
Population: All randomized participants receiving ≥1 dose of therapy and having MTT measurement either at Week 0 (BL) or end of Treatment Period 1. N=number of participants included in the Longitudinal Data Analysis (LDA) model
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 59 | 17 | 19 | 21 | 15
mg/dL | -5.2 (5.9) | -20.1 (10.3) | -25.6 (10.2) | -73.0 (9.3) | -54.6 (10.3)
Statistical Analysis 1: Comparison: Placebo (PLA) vs MK-3577 AM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.174, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -14.9, 90% CI 2-sided [-33.0 to 3.2]
Statistical Analysis 2: Comparison: Placebo (PLA) vs MK-3577 PM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.063, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -20.4, 90% CI 2-sided [-38.4 to -2.4]
Statistical Analysis 3: Comparison: Placebo (PLA) vs MK-3577 BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; [statistical method as in outcome 1, analysis 1]; LSM Difference = -78.1, 90% CI 2-sided [-96.4 to -59.8]
Statistical Analysis 4: Comparison: Placebo (PLA) vs METF BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA Model; [statistical method as in outcome 1, analysis 3]; LSM Difference = -49.4, 90% CI 2-sided [-66.9 to -31.8]

4. Secondary Outcome: Percentage Change From Baseline (BL) After 4-Week Treatment in Low-Density Lipoprotein C (LDL-C) Levels
Description: Blood samples were obtained from all participants to measure LDL-C levels at Week 0 (Baseline) and Week 4 of each treatment period (Week 4 Visit, Week 8 Visit, Week 12 Visit, and Week 16 Visit). For each visit, LDL-C was measured over 2 days. The average of duplicate measurements (when available) was used in the analysis.
Time Frame: Week 0 Visit (Baseline), Week 4 Visit, Week 8 Visit, Week 12 Visit, and Week 16 Visit
Population: All randomized participants who took at least 1 dose of study treatment and had a valid reading at timepoint.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage change from BL
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 102 | 100 | 99 | 86 | 18
percentage change from BL | 2.3 (25.0) [-1.6 to 6.3] | 1.5 (27.9) [-2.0 to 5.1] | 6.8 (27.9) [3.1 to 10.6] | 10.0 (21.8) [6.3 to 13.9] | -1.7 (23.4) [-7.7 to 4.8]
Statistical Analysis 1: Comparison: Placebo (PLA) vs MK-3577 AM; LDL-C values after log transformation were analyzed using a constrained LDA model that included terms for treatment, period, the interaction of treatment by period, prior antihyperglycemic therapy status (yes/no), and randomization stratum (participation in domiciled visits [yes/no]). Percentage change from baseline in LDL-C after 4-week treatment was reported, after back-transformation using the delta method with an alpha-level of 0.10 (2-sided); Test type: Superiority or Other; p = 0.742, LDA Model; LSM Difference = -0.8, 90% CI 2-sided [-4.6 to 3.1]
Statistical Analysis 2: Comparison: Placebo (PLA) vs MK-3577 PM; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.060, LDA Model; LSM Difference = 4.5, 90% CI 2-sided [0.6 to 8.4]
Statistical Analysis 3: Comparison: Placebo (PLA) vs MK-3577 BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, LDA Model; LSM Difference = 7.8, 90% CI 2-sided [3.8 to 11.7]
Statistical Analysis 4: Comparison: Placebo (PLA) vs METF BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.248, LDA Model; LSM Difference = -3.9, 90% CI 2-sided [-10.2 to 2.3]

5. Primary Outcome: Number of Participants With At Least One Adverse Event (AE) in the Treatment or Post-Treatment Periods
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the SPONSOR's product, is also an AE.
Time Frame: From first dose of study treatment (Week 0 Visit) to Week 18 Post-study Visit (up to 18 weeks).
Population: All randomized participants who took ≥1 dose of study treatment (N=118). Because this was a cross-over study, participants were counted in more than one treatment group. AEs were reported by the treatment that participants were receiving at the time of the event. Not all participants received all treatments.
Measure: Number; unit: Participants
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 108 | 106 | 105 | 89 | 18
Participants | 28 | 30 | 22 | 28 | 6

6. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 5
Time Frame: From first dose of study treatment (Week 0 Visit) to Week 16 Visit (up to 16 weeks).
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo (PLA) | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Number analyzed (Participants) | 108 | 106 | 105 | 89 | 18
Participants | 2 | 2 | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Week 0 Visit) to Week 18 Post-study Visit (up to 18 weeks).
Description: All randomized participants who took ≥1 dose of study treatment (N=118). Because this was a cross-over study, participants were counted in more than one treatment group. AEs were reported by the treatment that participants were receiving at the time of the event. Not all participants received all treatments.
Groups:
- Placebo: Participants received a placebo tablet matching the respective MK-3577 dose (10 mg, 6 mg, 25 mg) and metformin, depending upon randomization, for 4 weeks.
- MK-3577 AM: Participants received 10 mg MK-3577 orally QD in the AM for 4 weeks.
- MK-3577 PM: Participants received 6 mg MK-3577 orally QD in the PM for 4 weeks.
- MK-3577 BID: Participants received 25 mg MK-3577 orally BID for 4 weeks.
Arm/Group | Placebo | MK-3577 AM | MK-3577 PM | MK-3577 BID | METF BID
Serious Adverse Events (participants affected / at risk) | 1/108 | 2/106 | 2/105 | 0/89 | 0/18
Other Adverse Events (participants affected / at risk) | 3/108 | 4/106 | 3/105 | 5/89 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | MK-3577 AM (N=106) | MK-3577 PM (N=105) | MK-3577 BID (N=89) | METF BID (N=18)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | MK-3577 AM (N=106) | MK-3577 PM (N=105) | MK-3577 BID (N=89) | METF BID (N=18)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
A pre-specified interim analysis of the efficacy and safety data for the initial cohort of participants in this study (Cohort 1) determined that sufficient data had been accrued to assess the study hypotheses, thus the study was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR has the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.